CLINICAL TRIAL: NCT06815146
Title: Comparison of the Effects of Erector Spinae Area (ESP) Block and Mid-Transverse Process to Pleura Block(MTP) on Postoperative Opioid Consumption and Quality of Recovery in Lumbar Spinal Surgery
Brief Title: The Effects of ESP Block and Mid-Transverse Process to Pleura Block on Postoperative Opioid Consumption and Quality of Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, MD, Prof, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025
Record Dates: First submitted 2025-01-27; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Opioid Consumption; Quality of Recovery(QoR-40), Preoperative and Postoperative
Keywords: opioid consumption; quality of recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Blind patients and postoperative follow-ups will not know which group the patient is in the study. Randomization will be done with computer support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esp block (Active Comparator)
  Interventions: Diagnostic Test: Numeretic rating scale (NRS); Diagnostic Test: Quality of Results (QoR-40); Other: Opioid consuption
- mtp block (Experimental)
  Interventions: Diagnostic Test: Numeretic rating scale (NRS); Diagnostic Test: Quality of Results (QoR-40); Other: Opioid consuption

INTERVENTIONS:
Diagnostic Test: Numeretic rating scale (NRS) — NRS is a pain intensity determination system based on the person being asked to describe their pain on a scale of 0 (none), 10 (unbearable pain) and a point between.
Diagnostic Test: Quality of Results (QoR-40) — Several rating scales have been developed to measure quality of recovery after surgery and anaesthesia, but the most extensively used is the QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain.
Other: Opioid consuption — Opioid consuption will be recorded from PCA

SUMMARY:
Erector Spinae Area (ESP) Block and Mid-Transverse Process to Pleura Block(MTP) have recently been described for the treatment of pain after lumbar spinal surgery. Although these blocks have been shown to be effective in the treatment of pain after lumbar spinal surgery when compared with postoperative pain, they have not been compared in terms of the quality of recovery and opioid consumption after lumbar spinal surgery.

The aim of this clinical trial is to compare the effects of Erector Spinae Area (ESP) Block and Mid-Transverse Process to Pleura Block(MTP) on quality of recovery and opioid consumption in patients scheduled for lumbar spinal surgery. The effects of the 2 blocks on postoperative pain will also be compared and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elective Lumbar Spinal surgery performed
* ASA I-III
* 18-75 years old

Exclusion Criteria:

1. Refusal at enrollment
2. Request for withdrawal from the study
3. Inability to give informed consent
4. Emergency surgery
5. Bleeding diathesis
6. Presence of contraindications to the LA agents used in this study
7. Use of chronic opioids
8. Psychiatric disorders
9. Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | PCA results will be recorded at the 1st, 6th, 12th, 24th hours postoperatively.
  The patient will be administered tramadol PCA every eight hours and recorded.

SECONDARY OUTCOMES:
quality of recovery | 24 hours
  The quality of recovery (QoR-40) of patients who underwent both ESP block and MTP block at the 24th hour postoperatively will be evaluated with a scoring system.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eskin MB, Ceylan A, Ozhan MO, Atik B. Ultrasound-guided erector spinae block versus mid-transverse process to pleura block for postoperative analgesia in lumbar spinal surgery. Anaesthesist. 2020 Oct;69(10):742-750. doi: 10.1007/s00101-020-00848-w. Epub 2020 Sep 21. PMID 32955601